CLINICAL TRIAL: NCT06924034
Title: Early-phase Exercise-based Comprehensive Cardiac Rehabilitation Program After Myocardial Infarction: A Randomized Controlled Trial
Brief Title: Early-phase Exercise-based Cardiac Rehabilitation After MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ozge Ocaker Aktan, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06-07
Record Dates: First submitted 2025-03-30; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction (MI)
Keywords: Myocardial Infraction; MI; early phase; cardiac rehabilitation
MeSH Terms: conditions — Myocardial Infarction | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and Randomized Controlled experimental study. Participants were randomly divided into two groups in a 1:1 ratio; the study group and the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation Program (Experimental): Patients who perform Phase I and Phase II Cardiac Rehabilitation Program
  Interventions: Other: Phase I and Phase II Cardiac Rehabilitation Program
- Standard of care (No Intervention): The patients who received a usual care program

INTERVENTIONS:
Other: Phase I and Phase II Cardiac Rehabilitation Program — The program consisted of two stages: an inpatient phase lasting until discharge, followed by an outpatient-supervised Phase II lasting eight weeks. In the intervention group, the participants in the inpatient phase received active-participatory lower extremity movements and progressive walking training (i.e., progressive walking in the room-corridor-hospital) to prepare them for discharge. The inpatient phase I was conducted with supervision following the American Heart Association recommendations. Participants in the intervention group were then administered phase II of the supervised CR program. Phase II CR was performed 3 non-consecutive days a week for 8 weeks as an aerobic exercise program.
  Arms: Cardiac Rehabilitation Program

SUMMARY:
This study aimed to investigate the effects of early-phase exercise-based supervised cardiac rehabilitation on functional exercise capacity, grip strength, fatigue, sleep quality, and health-related quality of life.

DETAILED DESCRIPTION:
Myocardial infarction (MI) is not only a severe form of coronary heart disease but also a leading cause of death and physical disability, particularly in the rapidly growing elderly population. Although percutaneous coronary interventions reduce mortality, ensuring the recovery and reintegration of discharged patients into society remains an unresolved issue. Cardiac rehabilitation (CR) is beneficial for patients with MI in terms of reducing cardiovascular mortality and hospital readmissions, managing cardiovascular risk factors, and improving aerobic capacity.

CR is a comprehensive intervention tailored to the individual needs of patients diagnosed with heart disease. It includes personalized exercise training, physical activity promotion, health education, cardiovascular risk management, and psychological support. Initial recommendations for CR were limited to low-risk patients following MI. However, over the past two decades, with the accumulation of evidence supporting the benefits of CR, current clinical guidelines now routinely recommend comprehensive CR for a broader range of cardiac diagnoses, including acute coronary syndrome and heart failure with reduced ejection fraction.

Until two decades ago, studies recommended starting CR in the early phase, defined as the second-week post-discharge. However, in the past decade, CR initiation with very low-intensity exercise activity as early as one week after MI onset has been reported as safe and effective. More recently, studies have shown the beneficial effects of terminating bed rest within 12-24 hours and initiating bedside activities. Phase I exercise-based CR has been shown to be effective in improving exercise capacity and preventing recurrent cardiac events. Nonetheless, concerns remain regarding early exercise-based CR due to exercise-induced ischemia after acute MI. While the effects of early rehabilitation initiated post-MI have been investigated in the literature, sufficient evidence has yet to be established.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and medically stable patients with first MI
* Prescribed cardiac rehabilitation by a cardiologist
* Being between 30-65 years old
* having ejection fraction (EF) of more than 20% (i.e. EF≥ 20%)
* being volunteer to participate

Exclusion Criteria:

* having coronary artery bypass graft surgery
* Being diagnosed with chronic renal failure
* Presence of unstable angina
* Atrial fibrillation
* Severe and symptomatic aortic stenosis
* Presence of decompensated heart failure
* Exercise-induced myocardial ischemia,
* Pericardial disease,
* Moderate-to-severe valve disease
* COPD or asthma
* BMI > 40 kg/m2
* Orthopedic and neurological problems that prevent exercise

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | 8 weeks
  Functional exercise capacity assessment with 6-minute walk test distance as meters
Functional exercise capacity | 8 weeks
  Functional exercise capacity assessment with 30 s sit-stand test repetitions

SECONDARY OUTCOMES:
SF-12 Health releated Quality of Life questionnaire | 8 weeks
  Health-related Quality of Life was assessed with the SF-12 Health-related Quality of Life questionnaire (range: 0-100). Lower values on this questionnaire indicate worse symptoms
MacNew Heart Disease Health releated Quality of Life questionnaire | 8 weeks
  Disease-specific Health-related Quality of Life was assessed with the MacNew Heart Disease Health-related Quality of Life questionnaire (range: 1-7). Lower values on this questionnaire indicate worse symptoms.
Fatigue | 8 weeks
  Fatigue was assessed with Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale (range: 0-52). Lower values on this scale indicate worse symptoms.
sleep quality | 8 weeks
  Sleep quality was assessed with the Pittsburgh Sleep Quality Index (range: 0-21). Higher values on this scale indicate worse symptoms.
Grip strength | 8 weeks
  Hand grip strength with a hand dynamometer (Jamar® ,dynamometer / Promedics Ltd., Blackburn, Lancashire, UK)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Ozalevli, Prof., Study Director — Dokuz Eylul University; Özge Ocaker Aktan, PhD (c), Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] Sjolin I, Back M, Nilsson L, Schiopu A, Leosdottir M. Association between attending exercise-based cardiac rehabilitation and cardiovascular risk factors at one-year post myocardial infarction. PLoS One. 2020 May 11;15(5):e0232772. doi: 10.1371/journal.pone.0232772. eCollection 2020. PMID 32392231
- [Background] Taylor RS, Dalal HM, McDonagh STJ. The role of cardiac rehabilitation in improving cardiovascular outcomes. Nat Rev Cardiol. 2022 Mar;19(3):180-194. doi: 10.1038/s41569-021-00611-7. Epub 2021 Sep 16. PMID 34531576
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274
- [Background] Dalal HM, Zawada A, Jolly K, Moxham T, Taylor RS. Home based versus centre based cardiac rehabilitation: Cochrane systematic review and meta-analysis. BMJ. 2010 Jan 19;340:b5631. doi: 10.1136/bmj.b5631. PMID 20085991
- [Background] Peixoto TC, Begot I, Bolzan DW, Machado L, Reis MS, Papa V, Carvalho AC, Arena R, Gomes WJ, Guizilini S. Early exercise-based rehabilitation improves health-related quality of life and functional capacity after acute myocardial infarction: a randomized controlled trial. Can J Cardiol. 2015 Mar;31(3):308-13. doi: 10.1016/j.cjca.2014.11.014. Epub 2014 Dec 11. PMID 25633911